Clinical Trial No: NCT05438771

## The Effects of Ankaferd Hemostat on Preventing Oral Mucositis in Colorectal Cancer Patients Receiving Chemotherapy

**Introduction:** The purpose of oral care is to reduce the effect of oral microbial flora and prevent infection, pain, and bleeding associated with cancer treatment. New agents are introduced each day to be used in the prevention and treatment of mucositis in cancer treatment. One of those agents is the Ankaferd hemostat. Ankaferd hemostat has pleiotropic effects and anti-infective characteristics in tissue healing. The purpose of this study is to evaluate the effectiveness of the Ankaferd hemostat in the prevention of oral mucositis due to chemotherapy in adult patients diagnosed with colorectal cancer.

**Material and Method:** The study was designed as a randomized controlled experimental study to be conducted with patients who are recently diagnosed with colorectal cancer and will receive the first course of chemotherapy. Data were collected using the Performance Score and the Oral Mucositis Evaluation Scale.

**Findings:** There is a significant difference in the mucositis symptoms on days 7 and 15 after chemotherapy in the ankaferd hemostat and the bicarbonate group (p<0.05). In the binary logistic regression analysis, among the factors affecting the formation of mucositis on day 7, only neutrophil and TSH were included in the model, while only the TSH variable is statistically significant.

**Discussion and Conclusion:** A lower level of mucositis was found in the study compared to the other agents in the literature. It was determined that Ankaferd emostat is effective in preventing oral mucositis due to chemotherapy in adult patients diagnosed with colorectal cancer.